CLINICAL TRIAL: NCT00911794
Title: Pulmonary Therapy and Supplemental Written Disclosure Therapy for Chronic Lung Disease
Brief Title: Written Disclosure Therapy for Anxiety and Stress in Patients With Chronic Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Collaborators: Stony Wold-Herbert Fund, Inc. (Other)
Responsible Party: Adam Hurewitz M.D., Winthrop University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07300
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2009-06-02 (Estimated); Status verified 2009-06

CONDITIONS: Chronic Lung Diseases; COPD; Pulmonary Fibrosis
Keywords: Dyspnea; Written Disclosure Therapy; COPD; Pulmonary Fibrosis; Chronic Lung Diseases; Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Fibrosis; Dyspnea | interventions — salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Written Disclosure Therapy (Experimental)
  Interventions: Other: Disclosure Writing (Written Disclosure Therapy)
- Controls (Sham Comparator)
  Interventions: Other: Neutral (Sham) Writing

INTERVENTIONS:
Other: Disclosure Writing (Written Disclosure Therapy) — Patients write about a stressful life experience
  Other Names: Written Disclosure Therapy
  Arms: Written Disclosure Therapy
Other: Neutral (Sham) Writing — Patients write about neutral subjects
  Other Names: Sham Writing (Controls that wrote about neutral subjects)
  Arms: Controls

SUMMARY:
The purpose of this study is to determine whether Written Disclosure Therapy (WDT) is of any benefit to patients with chronic lung diseases who are participating in pulmonary rehabilitation.

DETAILED DESCRIPTION:
Chronic lung diseases are typically associated with impaired quality of life, stress, and anxiety. Written disclosure therapy (WDT) reduces stress in patients with a variety of chronic illnesses. We sought to determine if written disclosure therapy benefits patients with chronic lung diseases when it is added as a component to the pulmonary rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD or Pulmonary Fibrosis
* First time participants in Pulmonary Rehabilitation program

Exclusion Criteria:

* Dementia
* Prior significant psychiatric illness
* Inability to complete the questionnaires
* Inability cooperate with spirometry
* Inability or to participate in outpatient follow-up over the six-month

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Dyspnea and quality of life | Two-month and six-month time

SECONDARY OUTCOMES:
Six-minute walk distance | Two-month and six-month time
Spirometry values (FEV1 and FVC) | Two-month and six-month time

CONTACTS AND LOCATIONS:
Overall Officials: Adam Hurewitz, M.D., Principal Investigator — Winthrop University Hospital